CLINICAL TRIAL: NCT02699437
Title: Prevalence of Antiphospholipid Antibodies Among Women With Preeclampsia
Status: Completed | Type: Observational
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: HME
Record Dates: First submitted 2016-02-26; First posted 2016-03-04 (Estimated); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Antiphospholipid Antibodies
MeSH Terms: conditions — Pre-Eclampsia | interventions — Antibodies, Antiphospholipid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples will be tested for anticardiolipin antibodies and lupus anticoagulant
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women with preeclampsia: Testing for antiphospholipid antibodies (anticardiolipin antibodies and lupus anticoagulant) will be performed in pregnant women with preeclampsia.
  Interventions: Other: Testing for antiphospholipid antibodies

INTERVENTIONS:
Other: Testing for antiphospholipid antibodies — Blood samples will be tested for anticardiolipin antibodies and lupus anticoagulant

SUMMARY:
The purpose of this study is to determine the prevalence of positive antiphospholipid antibodies among women with preeclampsia and to determine the effect of antiphospholipid antibodies on the severity of preeclampsia and the obstetric outcomes

DETAILED DESCRIPTION:
For all women included in the study, blood samples will be tested for anticardiolipin antibodies and lupus anticoagulant. The clinical details of all women will be collected by reviewing their hospital and prenatal records. The following clinical characteristics will be evaluated: maternal age, previous gestations, parity, past or family history of preeclampsia, gestational age at the onset of preeclampsia, gestational age at delivery and birth weight. The following pregnancy and delivery complications will be assessed: placental insufficiency, intrauterine growth restriction, fetal loss (stillbirth) and early neonatal death.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with preeclampsia.

Exclusion Criteria:

* Women with systemic autoimmune disease.
* Women with active thromboembolic disorders.
* Women with history of previous thromboembolic disorders.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Attendants of Tertiary Hospital Obstetric Outpateint Clinics and Emergency Department
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of positive antiphospholipid antibodies | 20 weeks to 42 weeks gestational age
  Number of women having positive antiphospholipid antibodies per total number of women

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa M El-Shafiey, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University; Alaa El-Din M El-Gohary, Dr, Study Director — Mansoura University; El-Said M Abd El-Hady, Prof, Study Chair — Mansoura University
Locations (1):
- Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided